CLINICAL TRIAL: NCT04969978
Title: CONNECT: COmpreheNsive TraiNing and Engagement in Cessation Treatment
Brief Title: Electronic Quitline Referral With Enhanced Academic Detailing for the Promotion of Smoking Cessation
Acronym: CONNECT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Kaiser Permanente (Other); OCHIN, Inc. (Other); Oregon Health and Science University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steffani Bailey, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00023019; NCI-2021-06581 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00023019 (Other: OHSU Knight Cancer Institute); R01CA255016 (NIH)
Record Dates: First submitted 2021-07-09; First posted 2021-07-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Tobacco-Related Carcinoma; Smoking &Amp; Tobacco Cessation
MeSH Terms: conditions — Smoking; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Quitline eReferral) (Active Comparator): Clinics are notified via email that the Quitline eReferral system is available with a link to an online publication that includes an overview of Quitline services, information on Quitline effectiveness, and a detailed eReferral workflow with corresponding EHR screenshots, including how to identify eligible patients, create an eReferral, and access Quitline follow-up data in the EHR. Clinics also gain access to technological assistance, as needed.
  Interventions: Other: Informational Intervention
- ARM II (Quitline eReferral plus enhanced AD) (Experimental): Clinics receive standard online materials access to remote technological assistance as in Arm I. Clinics also receive group training of clinic staff prior to activation of the eReferral system and 12 months post-activation, follow-up booster sessions and monthly performance audit and feedback.
  Interventions: Behavioral: Enhanced Academic Detailing; Other: Informational Intervention

INTERVENTIONS:
Behavioral: Enhanced Academic Detailing — * Group training of clinic staff prior to activation of the eReferral system and 12 months post-activation
  * Follow-up booster sessions
  * Monthly performance audit and feedback
  Other Names: EAD
  Arms: ARM II (Quitline eReferral plus enhanced AD)
Other: Informational Intervention — Receive overview of Quitline services and use of Quitline eReferral via online materials

SUMMARY:
This phase IV clinical trial determines the impact of implementing a Quitline electronic (e)Referral system with an enhanced academic detailing implementation strategy on Quitline reach, tobacco cessation assistance and self-reported quit rates among patients in community health centers. It also examines the cost-effectiveness of Quitline eReferrals both with and without enhanced academic detailing. If this implementation strategy is effective, this strategy could be used to increase tobacco cessation treatment through the collaboration between state Quitlines and community health centers that serve large numbers of socioeconomically disadvantaged patients who use tobacco.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Implement a Quitline electronic (e)Referral system with enhanced academic detailing (AD) (intervention; n=10 community health centers [CHCs]) and without enhanced AD (comparison; n=10 CHCs) to compare rates of eReferral offers, eReferral acceptance, Quitline enrollment, orders for tobacco cessation medication, and receipt of in-clinic counseling among patients identified as currently using tobacco.

II. Assess the effectiveness of implementing a Quitline eReferral system with enhanced AD (intervention) versus without enhanced AD (comparison) on self-reported tobacco quit rates among all patients identified as current persons using tobacco using electronic health record (EHR) data.

III. Estimate the total annual costs and incremental cost-effectiveness of a Quitline eReferral system, with and without enhanced AD.

OUTLINE: Clinics are randomized to 1 of 2 arms.

ARM I: Clinics are notified via email that the eReferral system is available with a link to an online publication that includes an overview of Quitline services, information on Quitline effectiveness, and a detailed eReferral workflow with corresponding electronic health record (EHR) screenshots, including how to identify eligible patients, create an eReferral, and access Quitline follow-up data in the EHR. Clinics also gain access to technological assistance, as needed.

ARM II: Clinics receive standard online materials and access to remote technological assistance as in Arm I. Clinics also receive group training of clinic staff prior to activation of the Quitline eReferral system and 12 months post-activation, follow-up booster sessions and monthly performance audit and feedback.

ELIGIBILITY:
Study Clinic Inclusion Criteria:

* In Oregon
* On the OCHIN Epic EHR for >= 1 year
* Willing to be randomized to the intervention or comparison condition
* Willing to recruit a provider to serve as a clinic champion (to share monthly performance audit and feedback at all-staff meetings, determine desired content of booster sessions with clinic team members, and complete a survey at the completion of the intervention period) and a clinic manager to coordinate training and booster sessions

Study Patient Inclusion Criteria:

* Adult patients (>= 18 years of age)
* Identified as current tobacco users during >= 1 ambulatory and/or telehealth visit to one of the eligible study clinics over the 24-month study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9133 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2026-02-22 (Estimated)

PRIMARY OUTCOMES:
Accepted electronic (e)Referral to Quitline | At any point during the 24-month intervention period
  Proportion of patients who accepted a Quitline eReferral in intervention (EAD) versus comparator clinics. Will use a logistic mixed effects model that addresses the following design features of the study: 1) will include random intercept for clinic to account for clustering of patients within clinics; 2) will perform an intent-to-treat analysis; 3) hypothesis tests will be two-sided.

SECONDARY OUTCOMES:
Quitline eReferral offered | At any point during the 24-month intervention period
  Proportion of patients who were offered the Quitline eReferral in intervention (EAD) versus comparator clinics. Will construct similar logistic mixed effects models.
Quitline enrollment | At any point during the 24-month intervention period
  Proportion of patients who accepted the Quitline eReferral and enrolled in Quitline services in intervention (EAD) versus comparator clinics. Will construct similar logistic mixed effects models.
Receipt of in-office counseling | At any point during the 24-month intervention period
  Proportion of patients with an indication in the electronic health record (EHR) of receipt of counseling during an office visit in intervention (EAD) versus comparator clinics. Will construct similar logistic mixed effects models.
Tobacco cessation medication ordered | At any point during the 24-month intervention period
  Proportion of patients with a tobacco cessation medication in the 'medication orders' list of the EHR in intervention (EAD) versus comparator clinics. Will construct similar logistic mixed effects models.
Tobacco cessation | At any point during the 24-month intervention period or up to 6 months post-intervention
  Proportion of patients with EHR status change from current to former tobacco use. Will utilize similar generalized linear mixed model (GLMM) modeling to estimate the impact of the intervention on cessation outcomes.
Annual intervention costs | Years 1-4
  Mean total annual costs in years 1-4 to implement the eReferral into the EHR and maintain eReferral system, with and without enhanced academic detailing.
Cost-effectiveness | Years 1-4
  Mean total annual costs over years 1-4 by study arm, overall and for patients enrolled in the Quitline.
Incremental cost-effectiveness ratio | Years 1-4
  Difference in total costs by study arm, overall and for patients enrolled in Quitline.

OTHER OUTCOMES:
Tobacco use assessed | At any point during the 24-month intervention period
  Proportion of patients who had a current tobacco use assessment in intervention (EAD) versus comparator clinics.

CONTACTS AND LOCATIONS:
Overall Officials: Steffani Bailey, Principal Investigator — OHSU Department of Family Medicine
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Limited data set was given by partner research organization under data use agreement that excludes disclosure of any data outside of this study.